CLINICAL TRIAL: NCT03014778
Title: Efficacy Comparison of Two Vaginal Solutions for Preoperative Use in Candidate Women for Vaginal Surgeries
Brief Title: Efficacy of Two Vaginal Solutions in Preoperative Use
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Sharon Tzemach, Dr, HaEmek Medical Center, Israel
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 0093-15-EMC
Record Dates: First submitted 2017-01-04; First posted 2017-01-09 (Estimated); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Vaginal Surgeries
MeSH Terms: interventions — Povidone-Iodine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- The Chlorhexidine gluconate arm (Experimental): 35 women undergoing surgery will be vaginally pre-op washed by 0.05% chlorhexidine gluconate, 50 cc for 1 minute. 3 samples will be taken for culture: before, 10 minutes and 30 minutes after the wash.
  Interventions: Drug: The Chlorhexidine gluconate 0.05%
- The Povidone iodine arm (Active Comparator): 35 women undergoing surgery will be vaginally pre-op washed by 10% Povidone iodine, 50 cc for 1 minute. 3 samples will be taken for culture: before, 10 minutes and 30 minutes after the wash.
  Interventions: Drug: 10% Povidone iodine

INTERVENTIONS:
Drug: The Chlorhexidine gluconate 0.05% — Washing vagina pre- operatively with Chlorhexidine gluconate 0.05%
  Other Names: Sterets unisept
  Arms: The Chlorhexidine gluconate arm
Drug: 10% Povidone iodine — Washing vagina pre- operatively with 10% Povidone iodine
  Arms: The Povidone iodine arm

SUMMARY:
This study is necessary in order to provide proof the effectiveness of Chlorhexidine gluconate and its safety.

DETAILED DESCRIPTION:
It is well known from the literature that the use of Povidone-iodone based solution for vaginal preparation before surgery is fraught with side effects and sensitivity, and often does not provide sufficient eradication of colonies of pathogens from the operation field.

It is also known that Chlorhexidine gluconate in low concentration provides a better result and does not cause side effects more than Povidone-iodone, but the chlorhexidine is still not approved for washing the mucous membranes. This study is necessary in order to provide proof of its effectiveness and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Patients over the age of 18
2. Candidates for surgery (TOT- Trans Obturator Tape, cystoscopy, the introduction / removal of the stent the ureter, ureteroscopy), local or general anesthesia.

Exclusion Criteria:

1. A pregnant woman or post-partum.
2. A woman with known sensitivity to iodine, povidon or chlorhexidine.
3. Previous pelvic surgeries within three months from the surgery planned.
4. Patients taking antibiotics within one month from the surgery planned.
5. Immunological failure patients.
6. Patient unwilling to participate in the study.
7. Patients who require the appointment of a guardian condition
8. Women assigned to undergo a regular cystoscopy (no further action).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2017-01-01; Primary Completion 2018-12-31 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Changing in the number of colonies that grew at every stage | Before the washing, 10 minutes after washing, 30 minutes after washing.

SECONDARY OUTCOMES:
Signs of local irritation mucosa after each bathing preparations by looking at the mucosa, at the end of the clinical assessment. | 30 minutes after washing.
The appearance of signs of systemic allergic reactions after each bathing by looking at the mucosa, at the end of the clinical assessment. | Before the washing, 10 minutes after washing, 30 minutes after washing.

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Tzemah, MD, Principal Investigator — Haemek MC
Locations (1):
- Haemek Medical Center, Afula, Afula, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Darouiche RO, Wall MJ Jr, Itani KM, Otterson MF, Webb AL, Carrick MM, Miller HJ, Awad SS, Crosby CT, Mosier MC, Alsharif A, Berger DH. Chlorhexidine-Alcohol versus Povidone-Iodine for Surgical-Site Antisepsis. N Engl J Med. 2010 Jan 7;362(1):18-26. doi: 10.1056/NEJMoa0810988. PMID 20054046
- [Background] American College of Obstetricians and Gynecologists Women's Health Care Physicians; Committee on Gynecologic Practice. Committee Opinion No. 571: Solutions for surgical preparation of the vagina. Obstet Gynecol. 2013 Sep;122(3):718-20. doi: 10.1097/01.AOG.0000433982.36184.95. PMID 23963423
- [Background] Niedner R. Cytotoxicity and sensitization of povidone-iodine and other frequently used anti-infective agents. Dermatology. 1997;195 Suppl 2:89-92. doi: 10.1159/000246038. PMID 9403263
- [Background] Vorherr H, Vorherr UF, Mehta P, Ulrich JA, Messer RH. Vaginal absorption of povidone-iodine. JAMA. 1980 Dec 12;244(23):2628-9. PMID 7431610
- [Background] Kjolhede P, Halili S, Lofgren M. Vaginal cleansing and postoperative infectious morbidity in vaginal hysterectomy. A register study from the Swedish National Register for Gynecological Surgery. Acta Obstet Gynecol Scand. 2011 Jan;90(1):63-71. doi: 10.1111/j.1600-0412.2010.01023.x. Epub 2010 Nov 26. PMID 21275917
- [Background] Culligan PJ, Kubik K, Murphy M, Blackwell L, Snyder J. A randomized trial that compared povidone iodine and chlorhexidine as antiseptics for vaginal hysterectomy. Am J Obstet Gynecol. 2005 Feb;192(2):422-5. doi: 10.1016/j.ajog.2004.08.010. PMID 15695981